CLINICAL TRIAL: NCT01684098
Title: A Phase II Clinical Study to Evaluate the Safety and Efficacy of FalateScan (Technetium Tc 99m EC20) in Patients With Known Suspected Recurrent or Metastatic Cancer From a Solid Tumor
Brief Title: Safety and Efficacy of FalateScan (Technetium Tc 99m EC20) in Patients With Known Suspected Recurrent or Metastatic Cancer From a Solid Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.8
Record Dates: First submitted 2012-09-09; First posted 2012-09-12 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2012-09

CONDITIONS: Recurrent or Metastatic Cancer; Head and Neck Cancer; Pancreas Cancer; Bladder Cancer; Testicular Cancer
Keywords: recurrent or metastatic cancer; head and neck cancer; pancreas cancer; bladder cancer; testicular cancer
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Head and Neck Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Testicular Neoplasms

ARMS (1):
- Tc 99m EC20 (Other)
  Interventions: Drug: Tc 99m EC20

INTERVENTIONS:
Drug: Tc 99m EC20

SUMMARY:
The folate receptor is over-expressed on many types of cancer cells and new folate receptor targeted therapies are being developed to target cancer cells that over-express the folate receptor. As with other targeted therapies, it is important to develop diagnostic tests that will provide accurate information on folate receptor status and aid in selecting patients that may benefit from folate-targeted therapy.

DETAILED DESCRIPTION:
This Phase II, limited institution, open-label, single-arm, baseline-controlled study is designed to obtain data on the percentage of patients with recurrent or metastatic cancer from a solid tumor (including, but not limited to, breast, lung, mesothelioma, liver, colorectal, prostate, head and neck, pancreas, bladder and testicular cancer) with increased uptake of FalateScan in tumors, correlate the immunohistochemical staining findings with the FolateScan images, and verify product safety in patients with suspected recurrent or metastatic disease from any solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following eligibility requirements to be enrolled in the study:

  1. Patient must be 18 years of age or older.
  2. Patient must have known or strongly suspected recurrent or metastatic cancer from a solid tumor with at least one identifiable lesion > 1.5 cm as diagnosed by conventional imaging.
  3. Patient must have adequate kidney function defined as serum creatinine of < 1.5 X ULN.
  4. Patient must have adequate liver function defined as transaminases (SGOT and/or SGPT) may be up to 2.5 X ULN if alkaline phosphatase is <ULN or alkaline phosphatase may be up to 2.5 X ULN if Transaminases are < ULN. If alkaline phosphatase is outside of these parameters and is due to bone metastases verified by assessment of isoenzymes, then the subject is eligible.
  5. Patient must provide written informed consent prior to enrollment.

Exclusion Criteria:

* Patients must be excluded in any of the following conditions are present:

  1. Patient is pregnant or breastfeeding.
  2. Patient is simultaneously participating in another investigational drug study, excluding the follow-up phase.
  3. Patient has received an investigational agent within 7 days prior to enrollment.
  4. Patient is unable to tolerate conditions for radionuclide imaging.
  5. Patient has been administered another radiopharmaceutical that would interfere with the assessment of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-08; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Nelson M Oyesiku, MD, PhD, Principal Investigator — Emory University